CLINICAL TRIAL: NCT03314168
Title: Effects of Different Volumes of Combined Training on Neuromuscular Parameters of Women in Initial Treatment for Breast Cancer: A Randomized Controlled Trial
Brief Title: Adaptations to Breast Cancer and Exercise
Acronym: ABRACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: João Henkin (Other)
Collaborators: Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor-Investigator, João Henkin, Principal investigator, Federal University of Rio Grande do Sul
Organization: Federal University of Rio Grande do Sul (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 72983017.3.0000.5347
Record Dates: First submitted 2017-10-10; First posted 2017-10-19 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Combined training; Fatigue
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Patients who are randomized in control group will receive the usual care in their respective hospital.
  Interventions: Other: Control group
- Single-set group (Experimental): Patients who are randomized in Single-set (SS) group, will receive 12-week of combined training, twice a week, composed by 10 resistance exercises and 20-25 minutes aerobic exercise at 80-95% of the second ventilatory threshold heart rate in a cycle. One-single set will be performed per exercise at 60-80%1-RM, with 1-1,5min of rest between the exercises.
  Interventions: Other: Combined training
- Multiple-sets group (Experimental): Patients who are randomized in Multiples-set (MS) group, will receive 12-week of combined training, twice a week, composed by 10 resistance exercises and 20-25 minutes aerobic exercise at 80-95% of the second ventilatory threshold heart rate in a cycle. Regarding resistance exercises, three set will be performed per exercise at 60-80%1-RM, with 1-1,5min of rest between sets and the exercises.
  Interventions: Other: Combined training

INTERVENTIONS:
Other: Combined training — Resistance exercises performed with different volumes (i.e. one-single set and multiple-sets) and 20-25 minutes of aerobic exercise will be performed twice a week, during 12 weeks.
  Other Names: Concurrent training
  Arms: Multiple-sets group; Single-set group
Other: Control group — The usual care will be recommended to avoid systematic physical exercise for 3 months and will receive general clinical recommendations such as nutritional intake and lifestyle issues in their respective hospital.
  Arms: Control group

SUMMARY:
This study aims to investigate the effects of different volumes of combined training on fatigue, neuromuscular variables, morphological, cardiorespiratory capacity, functionality, and quality of life, in breast cancer (BCa) women undergoing primary treatment. Two thirds will be the intervention group that will perform combined training, while the other third will be the control group that will have physiotherapy sessions.

DETAILED DESCRIPTION:
Although chemotherapy and radiation are mainstream treatment modalities, patients will often experience treatment-related side effects such as impairments to the neuromuscular and cardiovascular systems and reduction in quality of life (QoL).To date, numerous positive effects on neuromuscular and aerobic parameters in response to resistance and aerobic training have been reported when both training modalities were simultaneously performed (i.e. combined training - COMB) in BCa patients. However, there is a lack of data regarding the prescription of this modality in BCa patients, as the necessary dose of resistance training for significant improve in fatigue, neuromuscular, and quality of life. In this sense, no previous studies investigate the effect of different volumes of resistance training in BCa patients, providing important informations about the prescription in this clinical population.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnostic at I and II stages;
* Adjuvant or neoadjuvant chemotherapy (≤50% of sessions completed);
* More than 18 years.

Exclusion Criteria:

* Current smoking
* Diabetic neuropathy;
* Hypertension uncontrolled;
* Heart failure;
* Clinical depression;
* Skeletal muscle impairment which not allow physical exercise.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2017-10-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular fatigue | Changes from baseline are assessed after the intervention (week 13)
  Fatigue will be assessed by Fatigue index in isokinetic device.
Subjective fatigue | Changes from baseline are assessed after the intervention (week 13)
  Fatigue will be assessed by Piper fatigue scale (PFS). The PFS in its current form is composed of 22 numerically scaled, "0" to "10" items (i.e. 0, none fatigue; 10, severe fatigue) that measure four dimensions of subjective fatigue: behavioral/severity (6 items; # 2-7); affective meaning (5 items: # 8-12); sensory (5 items: # 13-17); and cognitive/mood (6 items: # 18-23). These 22 items are used to calculate the four sub-scale/dimensional scores and the total fatigue scores.

SECONDARY OUTCOMES:
Body composition | Changes from baseline are assessed after the intervention (week 13)
  Body composition will be assessed by Dual-energy X-ray absorptiometry
Muscle thickness | Changes from baseline are assessed after the intervention (week 13)
  Muscle thickness will be assessed by ultrasound images of quadriceps femoris and biceps.
Echo intensity | Changes from baseline are assessed after the intervention (week 13)
  Echo intensity is a grey scale for analyze the image that ranging from 0 (black) to 255 (white), and will be assessed by ultrasound images of quadriceps femoris and biceps.
VO2máx | Changes from baseline are assessed after the intervention (week 13)
  VO2máx will be assessed by an incremental protocol in a cycle ergometer
Knee extension muscle strength | Changes from baseline are assessed after the intervention (week 13)
  Knee extension muscle strength will be assessed by a bilateral 1-repetition maximum, reported in Kg.
Unilateral vertical bench press muscle strength | Changes from baseline are assessed after the intervention (week 13)
  Unilateral vertical bench press muscle strength will be assessed by an unilateral 1-repetition maximum on both sides, reported in Kg.
Knee extension peak torque | Changes from baseline are assessed after the intervention (week 13)
  Knee extension peak torque will be assessed by maximal voluntary isometric contraction on the right side, in a isokinetic dynamometer.
Quality of life assessed by European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30+Br23 | Changes from baseline are assessed after the intervention (week 13)
  Quality of life will be assessed by European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30+Br23. The EORTIC is composed by 53 questions scaled "0" to "4", and "0" to "7". These 53 items are used to compute four domains (i.e. global, functions, symptoms, and BR23 functions).
Functional Performance: Timed-up and go test | Changes from baseline are assessed after the intervention (week 13)
  The timed-up-and-go requires an individual to stand up from a seated position in a chair, walk 2.44m, turn around a cone, walk back to the chair and sit down.
Functional performance: 5-repetitions Sit-to-stand test | Changes from baseline are assessed after the intervention (week 13)
  For the 5-repetition sit-to-stand test, participants are instructed to start the test in a seated position with arms folded across the chest. After the start command, participants stand up until full knees extension and then back to a seated position. The time is stopped when the participants touch the seat after five complete repetitions.
Functional performance: 30-seconds arm-curl | Changes from baseline are assessed after the intervention (week 13)
  The arm-curl test determines the maximal number of times a 2kg dumbbell can be lifted with the dominant arm through elbow flexion in 30 seconds. Participants start the test seated in a chair, with arms extended and forearm maintained in supinated position during full range of motion.
Functional Performance: Stair Climbing | Changes from baseline are assessed after the intervention (week 13)
  For the stair-climbing test, participants are instructed to climb a 10-step staircase without skip steps or using the handrail (except in need of balance to prevent falls

CONTACTS AND LOCATIONS:
Overall Officials: Ronei Pinto, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Hospital Moinhos de Vento, Pôrto Alegre
  - Universidade Federal do Rio Grande do Sul, Pôrto Alegre

REFERENCES:
- [Derived] Henkin JS, Rosa DD, Morelle AM, Caleffi M, Pinto SS, Pinto RS. Exercise volume load in women with breast cancer: Study protocol for the ABRACE randomized clinical trial. Contemp Clin Trials Commun. 2022 Dec 20;31:101053. doi: 10.1016/j.conctc.2022.101053. eCollection 2023 Feb. PMID 36589863